CLINICAL TRIAL: NCT07251933
Title: A Multi-national Real-world Outcomes and Treatment Patterns Study of Lanadelumab (Takhzyro) in Paediatric Patients With Hereditary Angioedema (TAHORA)
Brief Title: A Study of Lanadelumab in Children With Hereditary Angioedema (HAE) in Multiple Countries
Status: Not yet recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-743-4038
Record Dates: First submitted 2025-11-19; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Hereditary Angioedema (HAE)
Keywords: Drug Therapy
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with HAE-C1INH: Paediatric participants with HAE-C1INH who initiated long-term prophylaxis (LTP) treatment with lanadelumab within a routine clinical setting will be included.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is a non-interventional study.

SUMMARY:
HAE is a rare condition. It causes sudden swelling under the skin and inside the body, like in the belly, throat, or genitals. This swelling happens because of a temporary leak in blood vessels but does not cause itching or hives. HAE is classified based on the amount of a protein in the blood called C1 inhibitor (C1-INH): HAE with normal C1-INH levels and HAE with limited or insufficient C1-INH levels (C1-INH deficiency). This study will concentrate on children with HAE C1-INH deficiency who have received Takhzyro (Lanadelumab) as prophylactic treatment.

The main goal of the study is to assess how well lanadelumab works in children with HAE-C1INH deficiency in everyday life. This will be measured by checking how long children who receive lanadelumab will be free of HAE attacks.

Other goals are to understand how children with HAE-C1INH deficiency are being treated with lanadelumab, how well the treatment works for them, how safe it is and how often these children need to use healthcare services (like doctor visits, hospital stays, etc.) because of their condition.

The study will only look at data already existing in the participants' medical records. No treatment will be given as part of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is aged 2 to less than (<) 12 years at the time of lanadelumab initiation and is expected to have at least 6 months of follow-up information before turning 12.
2. Participant has physician-confirmed diagnosis of HAE-C1INH.
3. Participant initiated LTP with lanadelumab during the eligibility period.
4. Signed consent/assent (where required by local regulations).
5. Participant's medical record contains documentation of HAE attacks in the pre-index period and after lanadelumab initiation.

Exclusion Criteria:

1. Participant was enrolled in a therapeutic investigational drug (lanadelumab or other drug) or device trial at index date.
2. Participant with no documented HAE attacks in the 12 months prior to index date.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Paediatric participants who have been diagnosed with HAE-C1INH in Germany, France, United Kingdom (UK), Israel, Argentina and Serbia.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who are Free of HAE Attacks | Up to 13 months
  Percentage of participants who are free of HAE attacks will be reported. A HAE attack is defined as the symptoms or signs consistent with an attack in at least 1 of the following locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx).

SECONDARY OUTCOMES:
HAE Attack Rate of Participants | Up to 13 months
HAE Attack-free Rate of Participants Relative to Prior Treatment | Up to 13 months
Association Between Covariates of Interest and Attack Free Rate | Up to 13 months
  Association between covariates of interest (e.g., age, sex, family history) and attack-free rate will be determined. Associations between attack free rate and covariates of interest will be modelled, using generalized linear models.
Number of Participants With HAE Attack Based on Attack Severity | Up to 13 months
  Number of participants with HAE attack based on attack severity (mild, moderate, severe, unknown) will be reported.
Number of Participants With HAE Attack Based on Location | Up to 13 months
  Number of participants with HAE attack based on location (e.g. extremities, abdominal, facial, laryngeal or genital) will be reported.
Number of Participants with Treatment History Before use of Lanadelumab | Up to 13 months
  Number of participants with treatment history (type of treatment, duration of treatment, reason for start/ discontinuation/ switch) before use of lanadelumab will be reported.
Average Duration of Lanadelumab Treatment | Up to 13 months
  Average duration of lanadelumab treatment will be reported.
Number of Participants Characterized Based on Lanadelumab Treatment Patterns | Up to 13 months
  Number of participants based on lanadelumab treatment patterns (e.g. setting of administration, interval of administration changes/dose modifications, reasons for initiation/discontinuation and modifications) will be reported.
Number of Participants With Treatments Received Following Lanadelumab Discontinuation | Up to 13 months
  Number of participants with treatments (e.g. type of treatment, reason for selection) received following lanadelumab discontinuation will be evaluated.
Number of Participants With Healthcare Resource Utilization (HRU) Outcomes | Up to 13 months
  HRU outcomes will include number of healthcare professional (HCP) visits, number of emergency department (ED) visits, number of inpatient hospitalizations, number of participants with admission to and days spent in intensive care unit related to HAE-C1INH, and number of school days missed will be reported.
Duration of Hospital Stay in Days Related to HAE-C1INH Hospitalizations | Up to 13 months
  Length of hospital stay in days related to HAE-C1INH hospitalizations will be reported.
Percentage of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 13 months
Percentage of Participants With Injection Site Reactions | Up to 13 months
  Percentage of participants with injection site reactions will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/